CLINICAL TRIAL: NCT00966589
Title: Chronic Groin Pain and Sportsman Hernia of Athletes: Randomized Study Between Conservative Treatment and Laparoscopic Hernioplasty (TEP)
Brief Title: Surgical or Conservative Treatment of Sportsman Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Hannu Paajanen, Doctor, Kuopio University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5204519
Record Dates: First submitted 2009-08-21; First posted 2009-08-27 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2010-03

CONDITIONS: Groin Pain
Keywords: groin pain; sportsman hernia; osteitis pubis; laparoscopic surgery
MeSH Terms: interventions — tetraethylpyrazine; Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conservative treatment (Sham Comparator): physiotherapy
  Interventions: Procedure: laparoscopic hernioplasty (TEP)
- surgery (Active Comparator): laparoscopic hernioplasty (TEP)
  Interventions: Procedure: laparoscopic hernioplasty (TEP)

INTERVENTIONS:
Procedure: laparoscopic hernioplasty (TEP) — Insertion of polypropylene mesh behind pubic bone
  Other Names: laparoscopic surgery in groin pain; surgical treatment of sportsman hernia

SUMMARY:
Five to ten percent of athletes and physical active adults are suffering chronic groin pain. The most common diagnoses are adductor tendinitis, sportsman hernia and osteitis pubis. Sportsman hernia is not a real hernia in the groin, but overuse injury of the groin muscles and tendons. No evidence-based treatment of this disabling condition has been found so far. Experimental surgical treatments are based on various hernioplasties. Laparoscopic extraperitoneal hernioplasty (TEP) is a mini-invasive and effective method to heal sportsman hernia in non-randomized cohorts.

DETAILED DESCRIPTION:
This prospective randomized study investigates the effect of active conservative treatment (rest, physical treatment, corticosteroid injections, anti-inflammatory analgesics) versus surgery (laparoscopic TEP) on the healing of sportsman hernia. Diagnosis of sportsman hernia is always based on careful clinical examination and magnetic resonance imaging. 25 patients with sportsman hernia are randomized into conservative treatment and 25 patients in surgery. The duration of follow-up is 1 year. The main end-point of treatments is disappearing of chronic groin pain (visual analogue scale, entering to sports).

ELIGIBILITY:
Inclusion Criteria:

* severe groin pain lasting > 6 months
* sportsman hernia

Exclusion Criteria:

* other diagnosis ruled out by MRI and clinical examination

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Decrease of groin pain measured by visual analogue scale (VAS) | 1 year

SECONDARY OUTCOMES:
Return to sport activities | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hannu EK Paajanen, MD, PhD, Study Director — Central Hospital of Mikkeli, Finland
Locations (1):
- Hannu Paajanen, Mikkeli, Mikkeli, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuikka L, Hermunen H, Paajanen H. Effect of pubic bone marrow edema on recovery from endoscopic surgery for athletic pubalgia. Scand J Med Sci Sports. 2015 Feb;25(1):98-103. doi: 10.1111/sms.12158. Epub 2013 Dec 18. PMID 24350624
- See also: PMID: 15472551 [PubMed - indexed for MEDLINE] — http://www.ncbi.nlm.nih.gov/sites/entrez